CLINICAL TRIAL: NCT00562523
Title: A Phase I Dose Escalation Study With Sorafenib Administered Continuously in Combination With Docetaxel Administered Once Every Three Weeks in Patients With Advanced Solid Tumors.
Brief Title: Sorafenib/Docetaxel Dose Escalation Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Head Clinical Pharmacology, Bayer HealthCare Pharmaceuticals Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12438
Record Dates: First submitted 2007-11-21; First posted 2007-11-22 (Estimated); Last update posted 2013-05-23 (Estimated); Status verified 2013-05

CONDITIONS: Neoplasms
Keywords: Cancer; Docetaxel; Sorafenib
MeSH Terms: conditions — Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006)

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — Sorafenib 400mg by mouth daily in combination with docetaxel 60mg/m2 IV once every 3 weeks

SUMMARY:
The purpose of this study is to: 1.) Evaluate how your body reacts to sorafenib when taken daily (continuously) in combination with docetaxel given every 3 weeks, and to determine the safety of the two drugs together.2.) Measure your blood levels of sorafenib and docetaxel at specific times after taking the medications.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Advanced histological or cytological documentation of cancer
* At least one evaluable lesion
* ECOG Performance Status of 0 or 1
* No more than one prior chemotherapy regimen (prior adjuvant therapy, immunotherapy or hormone treatment are allowed and not restricted)
* Life expectancy of at least 12 weeks
* No previous exposure to docetaxel or sorafenib
* Adequate bone marrow, liver and renal function as assessed by the following:

  * Hemoglobin greater than or equal to 9.0 g/dL
  * Absolute neutrophil count (ANC) greater than or equal to 2,500/mm3
  * Platelet count greater than or equal to 100,000/mm3 Hepatic
  * Total Bilirubin less than or equal to ULN
  * AST, ALT and Alkaline Phosphatase less than 1.5x ULN.
  * PT-INR/PTT less than 1.5 x ULN (Patients who are being prophylactically anti coagulated with an agent such as coumadin or heparin will be allowed to participate provided that the INR less than 1.5. In addition, these patients must be monitored at appropriate intervals throughout study)
  * Serum creatinine less than or equal to 1.5 x upper limit of normal

Exclusion Criteria:

* Myocardial infarction or symptomatic coronary artery disease (severe or unstable angina) within 6 months prior to screening
* Active clinically serious infections (> Grade 2 NCI-CTCAE Version 3.0)
* Uncontrolled seizure disorder. Use of cytochrome P450 enzyme-inducing antiepileptic drugs (phenytoin, carbamazepine or phenobarbital) is not allowed
* Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management
* Known human immunodeficiency virus (HIV) infection or chronic hepatitis B or C
* Peripheral neuropathy > Grade 1
* Thrombotic or embolic events (such as transient ischemic attacks, myocardial infarction, pulmonary embolus), within 6 months prior to screening
* Major surgery, open biopsy or significant traumatic injury within 4 weeks of first study treatment
* Pregnant or breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-11; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To determine the safety, maximum tolerated dose and dose-limiting toxicities of oral sorafenib | 6 weeks

SECONDARY OUTCOMES:
To determine if there is a pharmacokinetic interaction between sorafenib and docetaxel when they are administered together | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- United States (2):
  - Tampa, Florida
  - Philadelphia, Pennsylvania